CLINICAL TRIAL: NCT07390656
Title: Effects of Intradialytic Resistance and Flexibility Exercises on Clinical Outcomes in Hemodialysis Patients: A Pilot Randomized Controlled Trial
Brief Title: Intradialytic Resistance and Flexibility Exercise in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek GİBYELİ GENEK (Other)
Responsible Party: Sponsor-Investigator, Dilek GİBYELİ GENEK, Principal Investigator, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HD-EX-2020
Record Dates: First submitted 2026-01-22; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hemodialysis
Keywords: Intradialytic exercise; Resistance exercise; Flexibility exercise; Quality of life; Clinical outcomes
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Participants were assigned to resistance exercise, flexibility exercise, or usual care groups and followed in parallel during the study period.
Masking Description: Due to the nature of the exercise interventions, masking was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Resistance Exercise (Experimental): Participants performed supervised resistance exercise during routine hemodialysis sessions. Exercises were conducted three times per week during the first two hours of dialysis over the study period.
  Interventions: Behavioral: Resistance Exercise
- Flexibility Exercise (Experimental): Participants performed supervised flexibility and stretching exercises during routine hemodialysis sessions. Exercises were conducted three times per week during the first two hours of dialysis over the study period.
  Interventions: Behavioral: Flexibility Exercise
- Usual Care (Control) (No Intervention): Participants received usual hemodialysis care without any structured exercise program during dialysis sessions.

INTERVENTIONS:
Behavioral: Resistance Exercise — A structured resistance exercise program performed during routine hemodialysis sessions under supervision.
  Arms: Resistance Exercise
Behavioral: Flexibility Exercise — A structured flexibility and stretching exercise program performed during routine hemodialysis sessions under supervision.
  Arms: Flexibility Exercise

SUMMARY:
This study examined whether different types of exercise performed during hemodialysis sessions affect patients' health and quality of life. Patients receiving regular hemodialysis were assigned to resistance exercise, flexibility exercise, or usual care during dialysis. Changes in health-related outcomes were evaluated before and after the exercise period.

DETAILED DESCRIPTION:
This single-center pilot study was conducted to explore the effects of exercise performed during hemodialysis on patients' health. Adult patients undergoing maintenance hemodialysis participated in one of three groups: resistance exercise, flexibility exercise, or usual care without exercise. The exercise programs were carried out during routine dialysis sessions under supervision.

Patients' clinical measurements and self-reported health outcomes were assessed at the start of the study and again after completion of the exercise period. The study was carried out between December 2020 and April 2021 following approval by the institutional ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Receiving maintenance hemodialysis for at least 3 months
* Stable clinical condition
* Ability to participate in exercise during hemodialysis sessions
* Provided written informed consent

Exclusion Criteria:

* Acute illness or unstable cardiovascular disease
* Severe musculoskeletal or neurological conditions limiting exercise
* Recent hospitalization
* Cognitive impairment preventing cooperation
* Participation in another structured exercise program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in dialysis adequacy assessed by Kt/V (urea) | From baseline to 12 weeks
  Change in dialysis adequacy measured by single-pool Kt/V (urea).
Change in dialysis adequacy assessed by urea reduction ratio (URR) | From baseline to 12 weeks
  Change in dialysis adequacy measured by urea reduction ratio (URR), expressed as a percentage

SECONDARY OUTCOMES:
Change in Short Form-36 (SF-36) Health-Related Quality of Life score | From baseline to 12 weeks
  Change in health-related quality of life assessed using the Short Form-36 Health Survey (SF-36), a validated 36-item questionnaire.
  SF-36 domain scores range from 0 to 100, with higher scores indicating better health-related quality of life.
Change in Beck Depression Inventory score | From baseline to 12 weeks
  Change in depressive symptoms assessed using the Beck Depression Inventory (BDI). Scores range from 0 to 63, with higher scores indicating more severe depressive symptoms.
Change in body mass index (BMI) | From baseline to 12 weeks
  Change in body mass index (BMI), calculated as weight in kilograms divided by height in meters squared (kg/m^2). Higher BMI indicates greater body mass relative to height.
Change in fat tissue index (FTI) | From baseline to 12 weeks
  Change in fat tissue index (FTI) assessed by bioelectrical impedance analysis (BIA), calculated from fat tissue mass (FTM) normalized to height squared (kg/m^2).
Change in lean tissue index (LTI) | From baseline to 12 weeks
  Change in lean tissue index (LTI) assessed by bioelectrical impedance analysis (BIA), calculated from lean tissue mass normalized to height squared (kg/m^2).
Change in physical function assessed by the 6-minute walk test (6MWT) | From baseline to 12 weeks
  Change in physical function assessed using the 6-minute walk test (6MWT), measured as the total distance walked in meters.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Gibyeli Genek, MD, Principal Investigator — Muğla Sıtkı Koçman University, Faculty of Medicine
Locations (1):
- Muğla Sıtkı Koçman University Training and Research Hospital, Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data from this study.